CLINICAL TRIAL: NCT00900042
Title: Cytogenetic and Flow Cytometric Analysis of : Renal Cell Carcinoma: A Companion Protocol to SWOG-8949
Brief Title: SWOG-9023, DNA Analysis of Tumor Tissue From Patients With Metastatic Kidney Cancer
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000502305; SWOG-9023 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Cytogenetic Analysis; Flow Cytometry

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor diagnostic tissue

INTERVENTIONS:
Genetic: DNA ploidy analysis
Genetic: DNA stability analysis
Genetic: chromosomal translocation analysis
Genetic: cytogenetic analysis
Other: flow cytometry
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: DNA analysis of tumor tissue may help doctors predict how well patients will respond to treatment.

PURPOSE: This laboratory study is analyzing the DNA in tumor tissue from patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if cytogenetic abnormalities can predict clinical outcome, in terms of response to treatment and survival, in patients with metastatic renal cell carcinoma registered to the nephrectomy arm (arm I) of SWOG-8949.
* Correlate cytogenetic abnormalities and DNA content analysis (DNA index and S-phase fraction) with clinical outcome.

OUTLINE: This is a partially prospective, partially retrospective, multicenter, companion study.

Paraffin-embedded tumor tissue specimens from patients enrolled in SWOG-8949 are evaluated by cytogenetic analysis (e.g., presence of trisomy and loss of Y chromosome) and flow cytometric analysis (e.g., presence of nondiploid cells and presence of abnormal proliferation index).

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of renal cell carcinoma

  * Any T, any N, M1 disease as specified in SWOG-8949
* Eligible for and registered on the nephrectomy arm* (arm I) of SWOG-8949 NOTE: *Patients must be registered on this study before undergoing nephrectomy on SWOG-8949

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 1993-07; Primary Completion 2002-12 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Number of successes per number of evaluable samples | up to 4 years after registration
  Success is defined as obtaining at least 10 analyzable metaphases.
Number of abnormalities per number of successes | up to 4 years after registration
  Abnormality is defined as at lease one clonal chromosomal abnormality.
Correlation of tumor response to treatment with the type and number of abnormalities | up to 4 years after registration
  Abnormality is defined as at lease one clonal chromosomal abnormality.
Correlation of time from diagnosis to development of metastatic disease with the type and number of abnormalities | up to 4 years after registration
  Abnormality is defined as at lease one clonal chromosomal abnormality.
Correlation of time from first diagnosis of metastatic disease until death with the type and number of abnormalities | up to 4 years after registration
  Abnormality is defined as at lease one clonal chromosomal abnormality.

CONTACTS AND LOCATIONS:
Overall Officials: Robert P. Whitehead, MD, Study Chair — University of Texas